CLINICAL TRIAL: NCT07114081
Title: Exploring Pre-operative Prediction of Pelvic Endometriosis, the Local Inflammatory Environment and Response to Surgical Treatment
Brief Title: EndometrioSis PRediction and Assessment of InflammaTion
Acronym: ESPRIT
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22/PR/0483
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic laparoscopy — Minimal access surgery to determine the presence of characteristic endometriosis lesions on visual inspection of the pelvis

SUMMARY:
The goal of this observational study is to develop a non-invasive predictive algorithm for a diagnosis of endometriosis in a group of symptomatic women attending for their first laparoscopic surgical procedure for symptoms that are suspicious for pelvic endometriosis and to understand the role of peripheral markers of inflammation in enhancing this diagnosis.

The main questions it aims to answer are:

Can a non-invasive quantitative algorithm ('Endometriosis Diagnostic Index') accurately predict the presence or absence of pelvic endometriosis? Is the peripheral inflammatory environment (for example, presence of inflammatory cytokines and chemokine) different between people with and without endometriosis?

ELIGIBILITY:
Inclusion Criteria:

• Consecutive female patients age 18-50 undergoing laparoscopy with the suspicion of endometriosis (as indicated by any recording in secondary care medical notes of endometriosis being a possible finding at laparoscopy; all those undergoing laparoscopy for sub-fertility (no conception after ≥6 months of trying, excluding confirmed male factor); or pelvic pain symptoms (dysmenorrhea; non-cyclical pelvic pain; dyspareunia; dyschezia) who is not otherwise excluded.

Exclusion Criteria:

* previous surgically confirmed endometriosis;
* postmenopausal status;
* laparoscopy for acute indication (ectopic; tubo-ovarian abscess; adnexal torsion);
* suspicion of malignancy;
* the sole indication of tubal sterilisation;
* the sole indication of myomectomy;
* pregnant or breastfeeding;
* significant medical co-morbidities including HIV and/or hepatitis B or C infection;
* where gynaecology is not the primary team undertaking surgery;
* unable to have transvaginal ultrasound (TVUSS);
* declines to take part in the study;
* patient unable to understand verbal or written information in English;
* lack of capacity to consent at the point of recruitment;
* known safeguarding issues.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Consecutive female patients age 18-50 undergoing gynaecological laparoscopic surgery at included institutions
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Endometriosis predictive model | 24 months
  Multiple logistic regression model of predictive variables

SECONDARY OUTCOMES:
Markers of inflammation | 24 months
  Cytokine multiplex for markers of inflammation in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
TBC